CLINICAL TRIAL: NCT02207543
Title: Assessment of Patient Satisfaction in Palliative Cancer When They Return Home After Hospitalization in Palliative Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of patients
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PALSATIS
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-03

CONDITIONS: Cancer; Palliative Care; Home
Keywords: Cancer; Palliative care; home
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medical telephonecontact (Experimental): Evaluations will be conducted by telephone 15 days after hospital discharge, 30 days and then every month until 6 months.
  Interventions: Other: Medical telephone contact

INTERVENTIONS:
Other: Medical telephone contact — Evaluations will be conducted by telephone 15 days after hospital discharge, 30 days and then every month until 6 months.

SUMMARY:
The proposed work is part of a multidisciplinary approach to continuity of care in the particular context of the palliative phase of cancer. In conducting this study, we would like to characterize, at the regional level, satisfaction with the care of patients and their families in their care home situations palliative cancer. This evaluation will be based on questionnaires adapted versions in French language satisfaction questionnaires recently validated for patients in palliative situation and supported home care.

It will also identify the challenges faced by both patients, caregivers attending physicians.

The evaluation of these elements is a prerequisite to propose ways of improving at a hospital palliative care for output relay and anticipate the coordination of care for optimal care of the patient at home, to meet the expectations of different stakeholders, or even prevent certain readmissions "avoidable".

DETAILED DESCRIPTION:
- Background and rationale of the research project Palliative care is defined, according to the French Society for Support and Palliative Care as acute care delivered in a comprehensive approach to the person with a serious illness, progressive or terminal. Their goal is to relieve physical pain and other symptoms, but also take into account the psychological, social and spiritual suffering. According to this definition, palliative care is interdisciplinary, cater to the patient as a person and his family, at home or in an institution and strive to preserve the best possible quality of life until death.

Very few studies on the quality of life for patients at end of life were conducted in France. Among them, the TRAPADO study is a prospective study to evaluate the quality of care, quality of life and impact on the environment in three parallel cohorts of cancer patients in palliative phase according to their choice of inpatient traditional in palliative care or home. The interim analysis of this study, was published in 2006 in the journal Bulletin of cancer: patients expressed a priority choice for the home; there was a marked alteration of the overall quality of life, as measured by the EORTC-QLQC30, no statistically significant difference between home and hospital; anxiety level was higher in the hospital. Relatives were satisfied with the care of the patient with a good perception of the family fabric and expressed a lower level of psychosocial distress at home. Nevertheless, the terminal readmissions were common with a large majority of hospital deaths.

More recently, Régis Aubry, in the framework of the National Observatory on End of Life (ONFV), has conducted an extensive field survey, published in March 2013, up to the caregivers who meet together near home but also health professionals involved in supporting patients at end of life. The report of this work highlights the importance of developing palliative care in the home including the intervention of specialized teams and coordination of teams working at home.

Indeed, in France, while 81% of the French would "spend their last moments at home" (FIFG, 2010), only 25.5% of deaths occur at home (ONFV, 2012).

Faced with this reality, we were asked to know what elements can explain this discrepancy between this reality and the desire of patients. This issue was the subject of a preliminary study, conducted in 2013 in Lower Normandy region. We chose to study the management of patients with cancer in palliative home situation by their GP after hospitalization Identified beds Palliative Care (LISP) Centre François Baclesse Caen: 19 of the 23 patients assessed, have expressed their willingness on the place of death to their GP, wanted to die at home. Nearly half (48%) of patients in our study died in the hospital. GPs interviewed reported that maintaining the homes of these patients had been facilitated by the relief of distressing symptoms and the establishment of aid.

This finding demonstrates that the GP can often not only coordinate the sometimes complex palliative situations, at home and that the intervention of specialized teams, interdisciplinary, is fundamental to maintaining a home in the best possible conditions.

But what about the patient felt about his quality of life at home? After collecting feedback from GPs Lower Normandy, we would like to continue this work. In this context, we propose a pilot study, single-center, to assess the satisfaction of patients and their families in home support palliative phase of cancer.

- Emerging nature of research topics covered: The proposed work is part of a multidisciplinary approach to continuity of care in the particular context of the palliative phase of cancer. In conducting this study, we would like to characterize, at the regional level, satisfaction with the care of patients and their families in their care home situations palliative cancer. This evaluation will be based on questionnaires adapted versions in French language satisfaction questionnaires recently validated for patients in palliative situation and supported home care.

It will also identify the challenges faced by both patients, caregivers attending physicians.

The evaluation of these elements is a prerequisite to propose ways of improving at a hospital palliative care for output relay and anticipate the coordination of care for optimal care of the patient at home, to meet the expectations of different stakeholders, or even prevent certain readmissions "avoidable".

- Degree of risk-taking and innovative scientific approach: The situation at the end of life patient palliative situation of cancer remains a research context underdeveloped. This study is based on the involvement of patients and their caregivers, at this stage of the disease to assess their satisfaction with care when returning home after a hospital palliative care. It proposes indeed used for this self-administered to patients and their caregivers questionnaires adapted questionnaires in French version of the research team CANHELP.

- Impact and potential consequences of the project: The proposed pilot study should document the satisfaction What patients in palliative situation of their cancer during their care at home, as well as those around them, at the regional level. The implementation of this project will also be used to validate the feasibility of involving these actors in the difficult context of the end of life, to understand their needs, difficulties and feelings regarding the effective care . Thereafter, it may be considered a larger study to complete these first results, before proposing ways to improve whose impact on satisfaction with care remain to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient (s) age (s) of 18 or more;
* Patient (s) reached (s) from cancer wholly palliative phase (estimated life expectancy of less than 3 months) in the judgment of the investigator;
* Patient (s) hospital (s) in palliative care and candidate for a return home;
* Patient (s) able to communicate with the investigator or his representative;
* Patient (s) have received clear information on the diagnosis and prognosis of their disease;
* Free and informed consent signed.

Exclusion Criteria:

* Patient (s) under guardianship or unable to give informed consent;
* Patient (s) whose cognitive functions can not be questioned.
* Patient (s) whose psychological distress does not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient care satisfaction | 15 days after their home return
  Evaluation of satisfaction with the care of patients in palliative phase of cancer 15 days after their home return after hospitalization in palliative care.

SECONDARY OUTCOMES:
Satisfaction of the primary caregiver | Satisfaction of the primary caregiver will be evaluated at day 15, months 1 to 6
  Evaluation of the satisfaction of the primary caregiver of maintaining the home of his relatives with cancer in palliative phase

OTHER OUTCOMES:
Patient quality of life | Patient quality of life will be evaluated at day 15, months 1 to 6
  Evaluation of the quality of life of patients at home over time.
The type and intensity of symptoms | The type and intensity of symptoms will be evaluated on day 15, months1 to 6
  Characterize the type and intensity of symptoms, physical and mental, and supported over time;

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine GRACH, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François Baclesse, Caen, France